CLINICAL TRIAL: NCT05727761
Title: Pioglitazone-Metformin Combination Treatment for High Risk Oral Preneoplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ENT-2022-31139
Record Dates: First submitted 2023-01-19; First posted 2023-02-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Oral Leukoplakia
Keywords: oral leukoplakia; oral cancer prevention; pioglitazone; metformin; precancerous oral lesion
MeSH Terms: conditions — Leukoplakia, Oral

STUDY DESIGN:
Intervention Model Description: Treatment with pioglitazone-metformin (15mg/500mg) twice a day for 12 weeks in 36 total high risk oral leukoplakia patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- oral leukoplakia patients (Experimental): 36 total high risk oral leukoplakia patients.
  Interventions: Drug: pioglitazone-metformin

INTERVENTIONS:
Drug: pioglitazone-metformin — Treatment with pioglitazone-metformin (15mg/500mg) twice a day for 12 weeks

SUMMARY:
This is a Phase IIa oral cavity leukoplakia study of pioglitazone 15mg and metformin 500mg BID for 12 weeks. The primary objective is to determine the clinical and histologic changes of leukoplakia from baseline following a 12 week course of twice daily pioglitazone-metformin. Outcomes are defined as are a reduction of the leukoplakia grade in > 50% of treated participants and a partial or complete clinical response defined as 50% or greater reduction in the sum of measured targeted lesions. In addition, participants who show clinical and histologic improvement should correlate with a significant reduction of Ki-67 proliferative indices in lesions of these participants as compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven hyperplasia in high risk anatomic areas (floor of mouth, mobile tongue, oropharynx). Hyperplasia or dysplasia of any grade in any erythroplakia lesion. Mild, moderate or severe dysplasia within the lesion at any site of the oral cavity or oropharynx.
* Must have objective evidence of oral leukoplakia that is measurable in 2 dimensions per RECIST. The lesion(s) may be clinically characterized by leukoplakia, erythroplakia, erythro/leukoplakia. Lesions may be located in the oral cavity or oropharynx. However, the index lesion must be located in an anatomic site accessible by punch biopsy and be a minimum of 4mm x 8 mm to permit a 4mm punch biopsy.
* Age 18 years or older at the time of consent.
* Evidence of adequate organ function within 14 days prior to Day 1
* Able to comply with treatment (i.e. able to swallow a tablet whole, not crushed) and complete a 12 week course of twice daily medication as required by this study in the opinion of the treating investigator.
* Body mass index (BMI) is ≥ 18.5.
* Sexually active persons of child-bearing potential agrees to use adequate contraception (a hormonal method that has been in continual use for a minimum of 3 months prior to the study screening visit, a barrier method, or abstinence) for the duration of study participation.
* Provides voluntary written consent prior to the performance of any research related activity.

Exclusion Criteria:

* Pregnant or breastfeeding or planning to become pregnant.
* A concurrent diagnosis of Type I or Type II diabetes that is being treated with insulin or an antidiabetic agent. Participants whose Type II diabetes is controlled with diet and/or exercise alone are eligible provided they meet all other eligibility criteria.
* Participant is taking another investigational agent (not approved by the FDA for any indication).
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to ACTOplus Met, pioglitazone or metformin.
* Any contraindication to biopsy - this study requires a 4 mm punch biopsy of a lesion and of nearby normal tissue prior to treatment and at the end of the 12 week treatment period.
* History of bladder cancer, including in situ bladder cancer.
* History of invasive cancer (other than non-melanoma skin cancer or cervical cancer in situ) active within 18 months prior to the baseline study visit. (Participants who have a history of cancer that was curatively treated without evidence of recurrence in the 18 months prior to the baseline study visit are considered eligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Clinical change in leukoplakia | after 12 weeks of intervention or at early termination.
  a partial or complete clinical response defined as 50% or greater reduction in the sum of measured targeted lesions
histologic change in leukoplakia | after 12 weeks of intervention or at early termination.
  reduction of the leukoplakia grade in > 50% of treated participants
Change in Ki-67 | After 12 weeks of intervention or at early termination
  Ki-67 proliferative indices in lesions

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ondrey, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - HealthPartners, Saint Paul, Minnesota

REFERENCES:
- [Derived] Gates JC, Abouyared M, Shnayder Y, Farwell DG, Day A, Alawi F, Moore M, Holcomb AJ, Birkeland A, Epstein J. Clinical Management Update of Oral Leukoplakia: A Review From the American Head and Neck Society Cancer Prevention Service. Head Neck. 2025 Feb;47(2):733-741. doi: 10.1002/hed.28013. Epub 2024 Nov 25. PMID 39584361